# **Informed Consent Form**

### Title:

"The Effect of Asymmetrical vs. Symmetrical High Flow Nasal Cannula on the Work of Breathing: A randomised cross-over study."

NCT number: not yet assigned

Unique Protocol ID: 16171/09.04.2024

Date 09.04.2024

#### **HELLENIC REPUBLIC**

## MINISTRY OF HEALTH & SOCIAL SOLIDARITY





#### **PULMONOLOGY CLINIC**

**DIRECTOR: Professor Konstantinos Gourgoulianis** 

# PATIENT CONSENT FORM FOR INVASIVE MEDICAL MEASUREMENT TO ASSESS WORK OF BREATHING

| 1. I, the undersigned: |
|-------------------------------------------------------------|
| Address: |
| Telephone: |
| 2. My doctor explained the following to me: |
| A) The nature and purpose of the procedure in general terms |
| B) The risks associated with the procedure |

| ••••• | |
|---|---|
| C) The | e alternative treatment options |
| ••••• | |
| ••••• | |
| 3. | I accept that during the procedure, unforeseen situations may require an |
| | additional or different procedure than what was previously explained to me. Therefore, I give my consent and request that the doctor and/or their associates |
| | perform any medical acts they deem necessary. This consent also includes |
| 4 | conditions that were unknown to the doctor at the time the procedure began. |
| 4. | I give / do not give my consent for the procedure or process to be photographed or videotaped, which may include parts of my body, for medical, scientific research, or |
| | educational purposes, provided that my identity is not disclosed through the images or |
| 5. | accompanying captions. For the advancement of medical education, I consent / do not consent to the |
| 6 | presence of observers in the area where the procedure will take place. |
| 6. | I acknowledge that the University General Hospital of Larissa may, at its discretion, retain and use or display for scientific research, therapeutic, or |
| | educational purposes any material or tissues taken from my body during my |
| 7. | hospitalization. I am aware that all blank spaces in this document were either filled in or crossed |
| ,. | out prior to my signing. |
| ••••• | ••••••••••••••••••••••••••••••••••••••• |

(The patient or person legally authorized to consent)

| DATE:/ Time: |
|----------------------|
| (Doctor's Signature) |